CLINICAL TRIAL: NCT03597178
Title: Contact Lens Insertion and Removal in a Senior Subject Demographic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CR-6289
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Results first posted 2019-08-12 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Visual Acuity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- senofilcon A (Experimental): Subjects that are of at least 60 years of age and non-habitual contact lens wearers will receive instructions to insert and remove a contact lens from each eye.
  Interventions: Device: senofilcon A

INTERVENTIONS:
Device: senofilcon A — ACUVUE OASYS® 1-DAY with HydraLuxe™ Technology

SUMMARY:
This will be a pilot, one-visit, open-label, non-dispensing study. Subjects will be given instructions and then attempt to insert and remove a contact lens in each eye.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Must be at least 60 years of age at the time of screening.
  4. The subject must have normal eyes (i.e., no ocular medications or infections of any type).
  5. The subject must have best corrected visual acuity (BCVA) of 20/30 or better in each eye.

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. A habitual and adapted wearer of contact lenses (have worn a contact lens at least one time in the past 5 years).
  2. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
  3. Any systemic disease, autoimmune disease, or use of medication that may interfere with contact lens wear.
  4. Any ocular infection.
  5. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
  6. Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
  7. History of binocular vision abnormality or strabismus.
  8. Any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g., HIV, by self-report).
  9. Suspicion of or recent history of alcohol or substance abuse.
  10. History of serious mental illness.
  11. History of seizures.
  12. Employee of investigational clinic (e.g., Investigator, Coordinator, Technician)
  13. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion
  14. Any Grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale
  15. Any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Pall, OD, MS, FAAO, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (1):
- VRC-East, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 16 subjects were enrolled into this study. Of those enrolled, 2 failed to meet all eligibility criteria. Of 14 dispensed subjects all completed the study.
Groups:
- Senofilcon A: Subjects that wore senofilcon A during the entire duration of the study
Period: Overall Study
Arm/Group | Senofilcon A
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Dispensed Subjects: All subjects dispensed a study lens.
Arm/Group | All Dispensed Subjects
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.3 (2.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Overall Success Rate of Insertion and Removal of a Contact Lens
Description: The subject attempted to insert a contact lens in each eye. The subject were allowed to voluntarily end the contact lens insertion activity at any time prior to the 20-minute time point. The time of insertion for each eye or the time of stopping the insertion process for each eye was recorded. Similarly, the time of removal for each lens or the time of stopping the removal process for each lens was recorded.
Time Frame: Lens insertion and Removal, up to 2-Hours
Population: All subjects who successfully ompleted all study visits and did not substanially deviate from the protocol as deterined by the trial cohort review committee prior to database lock.
Measure: Number; unit: Percentage of eyes
Units Other Than Participants: Eyes
Groups:
- Senofilcon A: Subjects that inserted and removed the senofilcon A lens.
Arm/Group | Senofilcon A
Number analyzed (Participants) | 14
Number analyzed (Eyes) | 28
Percentage of eyes | 85.7

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 1 day per subject.
Groups:
- Senofilcon A: Subjects that wore the senofilcon A during any in this study.
Arm/Group | Senofilcon A
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT03597178/Prot_SAP_000.pdf